CLINICAL TRIAL: NCT01814137
Title: A Randomised Trial Comparing Efficacy and Safety After Intensification With Either Insulin Aspart Once Daily as add-on or Changing to Basal Bolus Treatment With Insulin Degludec and Insulin Aspart in Subjects With Type 2 Diabetes Previously Treated With Insulin Degludec/Insulin Aspart Twice Daily (BOOST®: INTENSIFY BID)
Brief Title: A Randomised Trial Comparing Efficacy and Safety After Intensification With Either Insulin Aspart Once Daily as add-on or Changing to Basal Bolus Treatment With Insulin Degludec and Insulin Aspart in Subjects With Type 2 Diabetes Previously Treated With Insulin Degludec/Insulin Aspart Twice Daily
Acronym: BOOST®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-4003; 2012-003152-37 (EudraCT Number); U1111-1132-2674 (Other: WHO)
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; insulin degludec; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp BID + IAsp OD (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: insulin aspart
- IDeg OD + IAsp TID (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — For subcutaneous (s.c., under the skin) administration twice daily in combination with up to 2 oral antidiabetic drugs (OADs- dose and dosing frequency of OAD should remain unchanged).
  Arms: IDegAsp BID + IAsp OD
Drug: insulin degludec — For subcutaneous (s.c., under the skin) administration once daily in combination with up to 2 oral antidiabetic drugs (OADs- dose and dosing frequency of OAD should remain unchanged).
  Arms: IDeg OD + IAsp TID
Drug: insulin aspart — For subcutaneous (s.c., under the skin) administration once daily. Dose of IDegAsp and IAsp are individually adjusted.
  Arms: IDegAsp BID + IAsp OD
Drug: insulin aspart — For subcutaneous (s.c., under the skin) administration three times a day. Dose of IDeg and IAsp are individually adjusted.
  Arms: IDeg OD + IAsp TID

SUMMARY:
This trial is conducted globally. The aim of the trial is to compare efficacy of insulin degludec/insulin aspart (IDegAsp) twice daily (BID) + insulin aspart (IAsp) once daily (OD) versus basal bolus with insulin degludec (IDeg) OD + IAsp three times a day (TID) in controlling glycaemia by evaluating glycosylated haemoglobin (HbA1c). The trial is an extension to trial NN5401-3941 (NCT01680341).

ELIGIBILITY:
Inclusion Criteria:

* HbA1c equal to or above 7.0% measured after 26 weeks of treatment in NN5401-3941 (NCT01680341), by central laboratory

Exclusion Criteria:

* Uncontrolled or untreated severe hypertension defined as systolic blood pressure equal to or above 180 mmHg and/or diastolic blood pressure equal to or above 100 mmHg
* Impaired liver function, defined as alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) equal to or above 2.5 times upper limit of normal
* Impaired renal function defined as serum-creatinine equal to or above 125 micromol/L (equal to or above 1.4 mg/dL) for males and equal to or above 110 micromol/L (equal to or above 1.3 mg/dL) for females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (39):
- United States (25):
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Avon, Illinois
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Tacoma, Washington
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
- Algeria (3):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Tizi Ouzou
- Germany (5):
  - Novo Nordisk Investigational Site, Erdmannhausen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert
- Malaysia (2):
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Kuala Selangor
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Denizli
  - Novo Nordisk Investigational Site, Gaziantep
  - Novo Nordisk Investigational Site, Hatay
  - Novo Nordisk Investigational Site, Istanbul

REFERENCES:
- [Result] Bebakar WM, Chaykin L, Herslov ML, Rasmussen S. Intensification of IDegAsp Twice Daily (Adding Insulin Aspart vs. Switching To Basal-Bolus): Exploratory Randomized Trial in Type 2 Diabetes. Diabetes Ther. 2017 Feb;8(1):197-205. doi: 10.1007/s13300-016-0213-8. Epub 2016 Nov 16. PMID 27853981
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 20 sites in 4 countries as follows: Germany: 1 site; Malaysia: 2 sites; Turkey: 1 site; United States: 16 sites. The subjects in this trial were to continue from trial NN5401-3941 (NCT01680341).
Pre-assignment Details: Subjects who did not reach the HbA1c target < 7.0% on IDegAsp BID after 26 weeks of treatment in trial NN5401-3941 were enrolled in this trial.
Groups:
- IDegAsp BID + IAsp OD: Subjects randomised to insulin degludec/insulin aspart (IDegAsp) twice daily (BID) + insulin aspart (IAsp) once daily (OD) , at the discretion of the investigator, started the doses of IDegAsp at week 26 in trial NN5401-3941 with breakfast and main evening meal and added 4 units of IAsp at lunch. IDegAsp was administered subcutaneously (s.c.) by injection in the thigh, the upper arm (deltoid area) or the abdominal wall. The chosen area of injection had to be the same throughout the trial, with rotation within a given region recommended. IAsp was injected s.c. with the main meal OD, preferably into the abdominal wall in accordance with local labelling. Additional doses of IAsp were only allowed, if needed due to intercurrent illness. Titration (self-titration) of both IDegAsp and IAsp was done once weekly. Titration of IAsp could also be done based on carbohydrate counting but at the investigator's discretion. IAsp dose reduction had to be done based on the investigator's discretion.
- IDeg OD + IAsp TID: Subjects randomised to insulin degludec (IDeg) OD + IAsp thrice daily (TID) were, at the discretion of the investigator, to start with 70% of the total daily dose of IDegAsp taken at Week 26 in trial NN5401-3941 as IDeg OD and 30% as IAsp divided into 3 doses. IDeg was administered s.c. by injection in the thigh, the upper arm (deltoid area) or the abdominal wall and the chosen area of injection had to be the same throughout the trial. Rotation of injection sites within a given region was recommended. The OD injection time could be changed from day to day. IAsp was injected s.c. with the main meals TID, preferably into the abdominal wall in accordance with local labelling. Additional doses of IAsp were only allowed, if needed. Titration (self-titration) of IDeg and IAsp was performed once weekly. Titration of IAsp could also be done based on carbohydrate counting but at the investigator's discretion. IAsp dose reduction had to be done based on the investigator's discretion.
Period: Overall Study
Arm/Group | IDegAsp BID + IAsp OD | IDeg OD + IAsp TID
Started | 20 | 20
Completed | 15 | 15
Not Completed | 5 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Unclassified | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp BID + IAsp OD | IDeg OD + IAsp TID | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (8.0) | 56.9 (8.1) | 57.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 15 | 11 | 26
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.9 (0.7) | 7.7 (0.6) | 7.8 (0.7)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 7.3 (3.5) | 8.6 (2.8) | 7.9 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects and missing data was imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp BID + IAsp OD | IDeg OD + IAsp TID
Number analyzed (Participants) | 20 | 20
percentage of glycosylated haemoglobin | 0.05 (0.20) | -0.49 (0.19)

2. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: A treatment emergent adverse event was defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last dose of the trial product.
Time Frame: During 26 weeks of treatment
Population: Safety analysis set (SAS) included all subjects receiving at least one dose of the investigational product.
Measure: Number; unit: number of events
Arm/Group | IDegAsp BID + IAsp OD | IDeg OD + IAsp TID
Number analyzed (Participants) | 20 | 20
number of events | 33 | 45

3. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes
Description: Confirmed hypoglycaemic episodes were defined as episodes that are either:
  * severe (i.e., an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions) or
  * biochemically confirmed by a PG value of <3.1 mmol/L (56 mg/dL), with or without symptoms consistent with hypoglycaemia.
Time Frame: During 26 weeks of treatment
Population: The SAS included all subjects receiving at least one dose of the investigational product.
Measure: Number; unit: episodes
Arm/Group | IDegAsp BID + IAsp OD | IDeg OD + IAsp TID
Number analyzed (Participants) | 20 | 20
episodes | 54 | 95

4. Secondary Outcome: Number of Treatment Emergent Nocturnal (00:01-05:59) Confirmed Hypoglycaemic Episodes
Description: Hypoglycaemic episodes were defined as nocturnal if the time of onset was between 00:01 and 05:59 hours inclusive. Confirmed hypoglycaemic episodes were defined as severe hypoglycaemic episodes and/or a measured PG below 3.1 mmol/L (below 56 mg/dL).
Time Frame: During 26 weeks of treatment
Population: The SAS included all subjects receiving at least one dose of the investigational product.
Measure: Number; unit: episodes
Arm/Group | IDegAsp BID + IAsp OD | IDeg OD + IAsp TID
Number analyzed (Participants) | 20 | 20
episodes | 13 | 12

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG after 26 weeks of treatment. FPG was analysed on blood samples from fasting subjects which were analysed centrally.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. One subject in each arm did not have FPG values from week 0.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp BID + IAsp OD | IDeg OD + IAsp TID
Number analyzed (Participants) | 19 | 19
mmol/L | -0.80 (3.59) | -2.57 (2.73)

ADVERSE EVENTS:
Time Frame: Adverse events were captured on the onset date on or after the first day of exposure to randomised treatment and no later than the last day of randomised treatment.
Description: The SAS included all subjects receiving at least one dose of the investigational product.
Arm/Group | IDeg OD + IAsp TID | IDegAsp BID + IAsp OD
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/20
Other Adverse Events (participants affected / at risk) | 16/20 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD + IAsp TID (N=20) | IDegAsp BID + IAsp OD (N=20)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD + IAsp TID (N=20) | IDegAsp BID + IAsp OD (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 3 (3)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Retinal aneurysm (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 4 (6) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the highly selected trial population randomised in this trial (N=40), the results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.